CLINICAL TRIAL: NCT01699685
Title: A Multicenter, Randomized, Double-blind, Single-dose Study to Assess the Effect of the QAB149 and NVA237 Combination Versus QAB149 Alone on Inspiratory Capacity in Patients With Moderate or Severe COPD.
Brief Title: Swiss studY for the Treatment of COPD Patients With the Free combiNation of indacatERol and GlYcopyrroniumbromide.
Acronym: SYNERGY
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CNVA237ACH01; 2012-002362-13 (EudraCT Number)
Record Dates: First submitted 2012-09-28; First posted 2012-10-04 (Estimated); Results first posted 2016-02-09 (Estimated); Last update posted 2016-02-09 (Estimated); Status verified 2016-01

CONDITIONS: Chronic Obstructive Pulmonary Disease: COPD
Keywords: Moderate to severe COPD patients are included; NVA; QAB
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — indacaterol; Glycopyrrolate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sequence A (Placebo Comparator): Patients will inhale QAB149 (capsule form in blister packs) + Placebo via Novartis Concept 1 SDDPI
  Interventions: Drug: QAB149; Drug: Placebo
- Sequence B (Active Comparator): Patients will inhale QAB149 plus NVA237 (capsule form in blister packs) via Novartis Concept 1 SDDPI
  Interventions: Drug: QAB149; Drug: NVA237

INTERVENTIONS:
Drug: QAB149 — Capsule form in blister packs inhaled with the Novartis Concept 1 SDDPI
Drug: Placebo — Capsule form in blister packs inhaled with the Novartis Concept 1 SDDPI
  Arms: Sequence A
Drug: NVA237 — Capsule form in blister packs inhaled with the Novartis Concept 1 SDDPI
  Arms: Sequence B

SUMMARY:
The study purpose is to evaluate the effect of QAB149

* NVA237 vs. QAB149 on static lung hyperinflation.

DETAILED DESCRIPTION:
This is a multicenter, randomized, double-blinded, single-dose, cross-over, placebo-controlled study. The primary endpoint was chosen to demonstrate the superiority of a single-dose of the combined inhalation vs. the mono inhalation regarding the Inspiratory Capacity (IC) peak value. A total of 78 patients will be randomized to complete two visits with two single doses of treatment. Patients will be randomized in a cross-over manner. Treatment visits will be separated by a study medication wash-out period.Treatments will be administered in a blinded fashion.

The patients will be male and female patients, ≥40 years of age, with a documented diagnosis of moderate or severe COPD according to Global Initiative for Chronic Obstructive Lung Disease (GOLD) criteria and >10-pack years history of smoking, FEV1 <80% and ≥30% of the predicted normal value.

ELIGIBILITY:
Inclusion criteria:

* Male and female patients, ≥40 years of age, with a documented diagnosis of moderate or severe COPD according to Global Initiative for Chronic Obstructive Lung Disease (GOLD) criteria and >10-pack year history of smoking
* FEV1 <80% and ≥30% of the predicted normal value who have signed an informed consent form prior to the initiation of any study-related procedure

Exclusion criteria:

* No COPD exacerbations within 6 weeks prior to dosing
* No concomitant lung disease such as asthma
* Nno requirement for long term oxygen treatment or history of lung reduction surgery
* No medical conditions that would interfere with the performance of spirometry
* No other medical condition that in the opinion of the investigator may cause the patient to be unsuitable for completion of the study or place the patient at potential risk form being in the study e.g. uncontrolled hypertension or unstable ischemic heart disease.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2012-11; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Corinne Wild, PhD, Study Director — Novartis Pharmaceuticals; Corinne Wild, PhD, Study Chair — Novartis Pharmaceuticals; Martin Brutsche, Prof. Dr. med., Principal Investigator — Cantonal Hospital of St. Gallen
Locations (10):
- Switzerland (10):
  - Novartis Investigative Site, Faltigberg-Wald, Canton of Zurich
  - Novartis Investigative Site, Basel, Switzerland
  - Novartis Investigative Site, Locarno, Switzerland
  - Novartis Investigative Site, Barmelweid
  - Novartis Investigative Site, Bern
  - Novartis Investigative Site, Crans-Montana
  - Novartis Investigative Site, Lausanne
  - Novartis Investigative Site, Lugano
  - Novartis Investigative Site, Sankt Gallen
  - Novartis Investigative Site, Walenstadtberg

REFERENCES:
- [Derived] Salomon J, Stolz D, Domenighetti G, Frey JG, Turk AJ, Azzola A, Sigrist T, Fitting JW, Schmidt U, Geiser T, Wild C, Kostikas K, Clemens A, Brutsche M. Indacaterol and glycopyrronium versus indacaterol on body plethysmography measurements in COPD-a randomised controlled study. Respir Res. 2017 Jan 11;18(1):13. doi: 10.1186/s12931-016-0498-1. PMID 28077140

RESULTS

PARTICIPANT FLOW:
Groups:
- Sequence A: QAB149 (150μg puff) + placebo followed by QAB149 (150μg puff) + NVA237 (50μg puff)
- Sequence B: QAB149 (150μg puff) + NVA237 (50μg puff) followed by QAB149 (150μg puff) + placebo
Period: Period 1
Arm/Group | Sequence A | Sequence B
Started | 39 | 39
Safety Population | 39 | 38
Full Analysis Population (FAS) | 38 | 38
Completed | 36 | 36
Not Completed | 3 | 3
Not completed — Adverse Event | 1 | 1
Not completed — Medical or ethical, noncompliance | 2 | 0
Not completed — Other | 0 | 1
Not completed — Patient request | 0 | 1
Period: Period 2
Arm/Group | Sequence A | Sequence B
Started | 36 | 36
Completed | 35 | 36
Not Completed | 1 | 0
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Population: Demographic summary by treatment group (safety population, N = 77)
Groups:
- Total: Total of all reporting groups
Arm/Group | Sequence A | Sequence B | Total
Number analyzed (Participants) | 39 | 38 | 77
Age, Continuous [Mean (Standard Deviation); unit: Years] | 65.62 (9.247) | 64.18 (7.447) | 64.91 (8.383)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 17 | 31
  Male | 25 | 21 | 46

OUTCOME MEASURES:

1. Primary Outcome: Inspiratory Capacity (IC) Peak Value
Description: IC was measured with spirometry conducted according to internationally accepted standards. Peak IC was defined as the maximum IC of the mean at one of the post-dose measurements (30min, 60min, 120min, 180min and 240min).
Time Frame: Day (0) 30minutes, 1, 2, 3, and 4 hours; Day (6) 30 minutes, 1, 2, 3, and 4 hours
Population: Full analysis set (FAS) included all randomized patients who received at least one dose of study medication during at least one study period. Participants with observations after 4 hours were included in the analysis.
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | Sequence A | Sequence B
Number analyzed (Participants) | 38 | 38
Liters
  Day 0 (n=38, 38) | 2.87 (0.808) | 2.94 (0.777)
  Day 6 (n=36, 36) | 2.99 (0.856) | 2.85 (0.707)

2. Secondary Outcome: Forced Expiratory Volume in One Second (FEV1)
Description: FEV1 was measured with spirometry conducted according to internationally accepted standards. FEV1 was at 30, 60, 120, 180, and 240 minutes post-dose. Spirometry equipment and performance of spirometric testing had to be in accordance with standards as outlined in the American Thoracic Society for the Standardization of Spirometry recommendations. The spirometry equipment used during the study had to meet or exceed these minimal ATS recommendations
Time Frame: Day (0) 30minutes, 1, 2, 3, and 4 hours; Day (6) 30 minutes, 1, 2, 3, and 4 hours
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | Sequence A | Sequence B
Number analyzed (Participants) | 38 | 38
Liters
  Day (0) 30 min post-dose | 1.49 (0.442) | 1.57 (0.505)
  Day (0) 1 hour post-dose | 1.50 (0.440) | 1.60 (0.506)
  Day (0) 2 hour post-dose | 1.51 (0.437) | 1.60 (0.506)
  Day (0) 3 hour post-dose | 1.53 (0.430) | 1.59 (0.500)
  Day (0) 4 hour post-dose | 1.53 (0.434) | 1.60 (0.492)
  Day (6) 30 min post-dose | 1.59 (0.437) | 1.52 (0.473)
  Day (6) 1 hour post-dose | 1.63 (0.465) | 1.53 (0.463)
  Day (6) 2 hour post-dose | 1.66 (0.462) | 1.55 (0.476)
  Day (6) 3 hour post-dose | 1.65 (0.455) | 1.56 (0.470)
  Day (6) 4 hour post-dose | 1.64 (0.473) | 1.56 (0.459)

3. Secondary Outcome: Inspiratory Capacity (IC)
Description: During the 4 hours following inhalation of the study treatment, inspiratory capacity (IC) was measured with spirometry conducted according to internationally accepted standards. IC was measured at 30, 60, 120, 180, and 240 minutes post-dose
Time Frame: within 4h after dosing
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | Sequence A | Sequence B
Number analyzed (Participants) | 38 | 38
Liters
  Day (0) 30 min post-dose | 2.67 (0.771) | 2.75 (0.751)
  Day (0) 1 hour post-dose | 2.67 (0.799) | 2.79 (0.774)
  Day (0) 2 hour post-dose | 2.69 (0.803) | 2.71 (0.709)
  Day (0) 3 hour post-dose | 2.74 (0.811) | 2.69 (0.800)
  Day (0) 4 hour post-dose | 2.74 (0.823) | 2.74 (0.754)
  Day (6) 30 min post-dose | 2.79 (0.826) | 2.40 (0.724)
  Day (6) 1 hour post-dose | 2.80 (0.810) | 2.72 (0.759)
  Day (6) 2 hour post-dose | 2.86 (0.846) | 2.74 (0.689)
  Day (6) 3 hour post-dose | 2.83 (0.841) | 2.69 (0.719)
  Day (6) 4 hour post-dose | 2.85 (0.799) | 2.68 (0.699)

4. Secondary Outcome: Forced Volume Capacity (FVC)
Description: FVC was measured with spirometry conducted according to internationally accepted standards. Measurements were made 30, 60, 120, 180, and 240 minutes post-dose. The standardized AUC FEV1 was calculated as the sum of trapezoids divided by the length of time
Time Frame: Day (0) 30minutes, 1, 2, 3, and 4 hours; Day (6) 30 minutes, 1, 2, 3, and 4 hours
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | Sequence A | Sequence B
Number analyzed (Participants) | 38 | 38
Liters
  Day (0) 30 min post-dose | 2.98 (0.917) | 3.00 (0.839)
  Day (0) 1 hour post-dose | 3.00 (0.966) | 3.02 (0.846)
  Day (0) 2 hour post-dose | 3.01 (0.947) | 3.04 (0.862)
  Day (0) 3 hour post-dose | 3.08 (0.946) | 3.04 (0.872)
  Day (0) 4 hour post-dose | 3.07 (0.968) | 3.07 (0.852)
  Day (6) 30 min post-dose | 3.19 (1.002) | 2.96 (0.788)
  Day (6) 1 hour post-dose | 3.25 (1.047) | 2.97 (0.807)
  Day (6) 2 hour post-dose | 3.29 (1.018) | 2.99 (0.754)
  Day (6) 3 hour post-dose | 3.32 (1.003) | 2.98 (0.794)
  Day (6) 4 hour post-dose | 3.30 (1.012) | 2.96 (0.797)

5. Secondary Outcome: Total Lung Capacity (TLC)
Description: TLC was measured with spirometry conducted according to internationally accepted standards. Peak TLC was calculated as the mean of the three Functional Residual Capacity peak measurements plus the mean of the three Inspiratory Capacity measurements which were measured each at 30, 60, 120, 180 and 240 minutes post dose
Time Frame: Day (0) 30minutes, 1, 2, 3, and 4 hours; Day (6) 30 minutes, 1, 2, 3, and 4 hours
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | Sequence A | Sequence B
Number analyzed (Participants) | 38 | 38
Liters
  Day (0) 30 min post-dose | 7.20 (1.587) | 6.81 (1.144)
  Day (0) 1 hour post-dose | 7.17 (1.559) | 6.79 (1.197)
  Day (0) 2 hour post-dose | 7.06 (1.658) | 6.81 (1.190)
  Day (0) 3 hour post-dose | 7.14 (1.662) | 6.82 (1.198)
  Day (0) 4 hour post-dose | 7.21 (1.608) | 6.78 (1.247)
  Day (6) 30 min post-dose | 7.20 (1.664) | 6.79 (1.243)
  Day (6) 1 hour post-dose | 7.12 (1.576) | 6.80 (1.312)
  Day (6) 2 hour post-dose | 7.21 (1.641) | 6.80 (1.213)
  Day (6) 3 hour post-dose | 7.23 (1.561) | 6.81 (1.304)
  Day (6) 4 hour post-dose | 7.30 (1.691) | 6.93 (1.376)

6. Secondary Outcome: Airway Resistance (Raw)
Description: Raw was measured with spirometry conducted according to internationally accepted standards. Raw was the mean of the measurements which were measured each at 30, 60, 120, 180 and 240 minutes
Time Frame: Day (0) 30minutes, 1, 2, 3, and 4 hours; Day (6) 30 minutes, 1, 2, 3, and 4 hours
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: cmH2O/l/s
Arm/Group | Sequence A | Sequence B
Number analyzed (Participants) | 38 | 38
cmH2O/l/s
  Day (0) 30 min post-dose | 5.13 (2.243) | 4.74 (1.810)
  Day (0) 1 hour post-dose | 5.19 (2.561) | 4.61 (1.881)
  Day (0) 2 hour post-dose | 5.21 (2.496) | 4.43 (1.849)
  Day (0) 3 hour post-dose | 5.07 (2.528) | 4.53 (1.748)
  Day (0) 4 hour post-dose | 5.18 (2.535) | 4.48 (1.866)
  Day (6) 30 min post-dose | 4.73 (2.540) | 5.18 (2.130)
  Day (6) 1 hour post-dose | 4.47 (2.323) | 4.97 (1.861)
  Day (6) 2 hour post-dose | 4.31 (2.119) | 4.71 (1.822)
  Day (6) 3 hour post-dose | 4.30 (2.161) | 4.77 (1.989)
  Day (6) 4 hour post-dose | 4.30 (2.170) | 4.78 (1.939)

ADVERSE EVENTS:
Arm/Group | Sequence A | Sequence B
Serious Adverse Events (participants affected / at risk) | 0/39 | 0/38
Other Adverse Events (participants affected / at risk) | 5/39 | 3/38
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Sequence A (N=39) | Sequence B (N=38)
Nasopharyngitis (Infections and infestations) | 1 | 0
Forced expiratory volume decreased (Investigations) | 1 | 1
Inspiratory capacity decreased (Investigations) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety.